CLINICAL TRIAL: NCT04151433
Title: BLAST: a Randomized Controlled Trial on Conservative Endometrioma Surgery Using the CO2 Laser: the Combined Technique Versus CO2 Laser Vaporization Only
Brief Title: Conservative Endometrioma Surgery
Acronym: BLAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: GZA Ziekenhuizen Campus Sint-Augustinus (Other); Centre Hospitalier Régional de la Citadelle (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S62899
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Endometriosis Ovary; Endometrioma
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The combined technique (Active Comparator): First step consisting of stripping the cyst wall for 80% of the surface, followed by a second step consisting of ablation of the remaining 20% cyst surface.
  Interventions: Procedure: Comparison between 2 different laparoscopic techniques in conservative surgical treatment of endometriomas (both arms are existing and accepted surgical strategies).
- CO2 laser vaporization only (Active Comparator): CO2 laser vaporization only of the complete inner cystic wall after drainage of the cyst content, irrigation and inspection of its inner wall. Ablation of the inner cyst wall using the CO2 laser (Lumenis). Power settings of 30-55W for CO2 laser beam and 6-10W for CO2 fibre are used. The laser should be on the ablate function to widen the beam (e.g. Surgitouch modus). The laser should be applied in Surgitouch modus so that it can ablate the cyst surface while preserving the underlying healthy tissue.
  Interventions: Procedure: Comparison between 2 different laparoscopic techniques in conservative surgical treatment of endometriomas (both arms are existing and accepted surgical strategies).

INTERVENTIONS:
Procedure: Comparison between 2 different laparoscopic techniques in conservative surgical treatment of endometriomas (both arms are existing and accepted surgical strategies). — cf. different arms

SUMMARY:
To study which surgical technique offers better results in treating endometriomas in terms of ovarian reserve preservation.

The 2 conservatives techniques used are:

1. The combined technique
2. CO2 laser vaporization only

Ovarian reserve will be assessed by consecutive measurements of AMH serum levels before and after surgery.

ELIGIBILITY:
Population: patients planned for laparoscopic CO2 laser surgery for endometriotic cysts.

Inclusion Criteria:

* Age: 18 - 40 years (both inclusive)
* Unilateral endometriotic cysts with a mean diameter of >=2.5cm and ≤8 cm, measured in 3 dimensions.
* Presence of a contralateral endometrioma of ≤ 2cm is allowed
* Complaining of infertility and/or pain
* BMI ≤35
* Use of contraception (combined or Progesteron only) for at least 4 weeks before surgery

Exclusion Criteria:

* Incomplete surgery for the pelvis
* Contra-indication for the use of contraception (combined or Progesteron only)
* Use of GnRH analogues preoperatively and in the first 3 months postoperatively
* (History of) hysterectomy
* Prior unilateral oophorectomy
* Pituitary/hypothalamic disorders
* Suspected malignancy
* Contralateral endometrioma of >2 cm
* AMH <0.7 preoperatively
* Pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
AMH levels 3 months postoperatively | 3 months postoperatively
  To assess the effect of conservative laparoscopic treatment of endometrioma(s) on ovarian reserve as reflected by AMH in patients planned for laparoscopic CO2 laser surgery. For the primary outcome evaluation of serum AMH will be done before (baseline) and after (at 3 months follow up) laparoscopic treatment of endometrioma(s).

CONTACTS AND LOCATIONS:
Overall Officials: Carla Tomassetti, MD, PhD, Principal Investigator — Leuven University Fertility Center
Locations (4):
- Belgium (4):
  - GZA Sint-Augustinus, Antwerp
  - Cliniques universitaires Saint-LUC (UCL), Brussels
  - UZLeuven, Leuven
  - CHR La Citadelle, Liège

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bafort C, Lie Fong S, Fieuws S, Geysenbergh B, Nisolle M, Squifflet JL, Tebache L, Wyns C, Meuleman C, Tomassetti C. Conservative endometrioma surgery: The combined technique versus CO2-laser vaporization only (BLAST: Belgium LAser STudy): Clinical protocol for a multicenter randomized controlled trial. PLoS One. 2025 Mar 6;20(3):e0315709. doi: 10.1371/journal.pone.0315709. eCollection 2025. PMID 40048474